CLINICAL TRIAL: NCT06938295
Title: Comparing Diagnostic Accuracy of High-End Intestinal Ultrasound Versus Mid-End Ultrasound With Tandem Ileo-Colonoscopy in Inflammatory Bowel Disease (The HUMID Study): A Paired, Validating Confirmatory Study
Brief Title: Comparing Diagnostic Accuracy of High-end Intestinal Ultrasound Versus Mid-end Ultrasound With Tandem Ileo-colonoscopy in Inflammatory Bowel Disease : a Paired, Validating Confirmatory Study
Acronym: HUMID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AIG/IEC-BH&R 61/09.2024-01
Record Dates: First submitted 2024-11-21; First posted 2025-04-22 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Ultrasound; Inflammatory bowel disease; Crohn's disease; Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult patients with inflammatory bowel disease (Active Comparator): Participants will undergo intestinal ultrasound (IUS) assessments using both a high-end (Samsung RS85) and a mid-end (Siemens ACUSON S2000) ultrasound machine to evaluate ileocolonic inflammation in inflammatory bowel disease (IBD). Each device is used within the same session, focusing on bowel wall thickness, vascularity, and structural changes. The high-end ultrasound provides advanced imaging capabilities, while the mid-end device offers standard IUS functionalities. Tandem ileo-colonoscopy is performed as the reference standard to validate findings.
  Primary Outcome: Diagnostic accuracy (sensitivity, specificity) of high-end vs. mid-end ultrasound.
  Secondary Outcome: Impact of ultrasound findings on clinical management decisions, evaluating cost-effective options for routine IBD monitoring.
  Interventions: Diagnostic Test: Comparative Use of High-End and Mid-End Intestinal Ultrasound Devices for IBD Disease activity assessment

INTERVENTIONS:
Diagnostic Test: Comparative Use of High-End and Mid-End Intestinal Ultrasound Devices for IBD Disease activity assessment — This study compares two intestinal ultrasound (IUS) devices-a high-end machine (Samsung RS85) and a mid-end machine (Siemens ACUSON S2000)-for assessing ileocolonic inflammation in IBD patients. The high-end device offers advanced imaging features, including high-resolution, speckle reduction, and extended field of view, allowing for detailed visualization of the bowel wall and vascularity. The mid-end device, while more basic, provides essential IUS functions for examining bowel wall thickness, structure, and inflammation markers. Both devices are used in a single clinical session, with results compared against tandem ileo-colonoscopy as the reference standard. This unique dual approach enables evaluation of the diagnostic performance of each device type. If comparable, the mid-end device may offer a cost-effective solution, increasing access to routine IUS in various healthcare settings, especially where high-end technology is limited.

SUMMARY:
The HUMID Study (High-end vs. Mid-end Ultrasound in IBD Diagnostics) is a prospective, cross-sectional, paired diagnostic accuracy study evaluating the performance of mid-end versus high-end intestinal ultrasound (IUS) machines in assessing ileocolonic involvement in patients with inflammatory bowel disease (IBD). Conducted at the Asian Institute of Gastroenterology, this study compares the Siemens ACUSON S2000 (mid-end) with the Samsung RS85 (high-end) ultrasound machines, using ileo-colonoscopy as the reference standard. All enrolled patients will undergo clinical evaluation, IUS with both machines, and colonoscopy. The primary objective is to assess and compare the diagnostic accuracy (sensitivity, specificity, PPV, NPV) of the two ultrasound systems. Secondary objectives include evaluating the impact of IUS findings on clinical management. The study aims to provide evidence for cost-effective imaging strategies in resource-limited settings where access to advanced diagnostics is restricted.

DETAILED DESCRIPTION:
The HUMID Study (High-end versus Mid-end Ultrasound in Inflammatory Bowel Disease Diagnostics) is a prospective, cross-sectional, paired diagnostic accuracy study designed to compare the performance of two intestinal ultrasound systems-a high-end system (Samsung RS85) and a mid-end system (Siemens ACUSON S2000)-in detecting ileocolonic inflammation in patients with inflammatory bowel disease. The study uses ileo-colonoscopy as the diagnostic reference standard and also evaluates the impact of ultrasound findings on clinical management and potential cost savings in resource-limited settings.

Eligible patients with known inflammatory bowel disease involving the colon and/or terminal ileum will undergo two intestinal ultrasound examinations followed by ileo-colonoscopy. To minimize operator bias, the mid-end ultrasound examination will be performed and interpreted by an experienced gastrointestinal sonologist using the Siemens ACUSON S2000 system. The high-end ultrasound examination will be conducted independently by an inflammatory bowel disease specialist using the Samsung RS85 system. Both sonographers will be blinded to each other's findings and to colonoscopy results. The examinations will be conducted in close succession on the same day, using standardized scanning protocols and probe frequencies suitable for bowel wall assessment.

Ultrasound assessments will include bowel wall thickness, mural stratification, vascularity, and disease extent. All findings will be recorded on pre-specified case report forms. Ileo-colonoscopy will be performed within 24 hours of the ultrasound exams by a separate blinded endoscopist. Endoscopic activity scores will be used as the reference standard for determining diagnostic accuracy.

The primary objective is to compare the diagnostic accuracy-measured by sensitivity, specificity, positive predictive value, and negative predictive value-of mid-end versus high-end ultrasound systems in detecting ileocolonic disease activity. The study aims to determine whether mid-end machines, which are more affordable and accessible, can offer comparable diagnostic performance to high-end systems.

Secondary objectives include assessing whether ultrasound findings lead to changes in clinical management. To ensure objectivity, an independent panel of three experienced inflammatory bowel disease physicians-blinded to the identity of the ultrasound machine-will review each case and determine whether ultrasound findings would have justified changes such as treatment escalation or de-escalation, surgical referral, or additional diagnostic evaluation. Panel decisions will be based on standardized clinical scenarios and will be adjudicated by consensus.

The study also includes a health-economic component, analyzing how the integration of mid-end ultrasound into clinical workflows may reduce reliance on invasive and high-cost diagnostics like colonoscopy or cross-sectional imaging. Real-world cost estimates will be used to model the economic impact.

By providing comparative data on diagnostic accuracy, management impact, and economic value, the HUMID Study seeks to inform clinical practice guidelines and promote the use of scalable ultrasound solutions in inflammatory bowel disease, particularly in resource-constrained healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years.
* Confirmed diagnosis of inflammatory bowel disease (IBD), specifically with ileocolonic involvement.
* Clinically stable at the time of assessment.
* Willing and able to undergo both intestinal ultrasound (IUS) assessments (mid-end and high-end) and the reference standard ileo-colonoscopy.
* Provides informed consent to participate in the study.

Exclusion Criteria:

* Pregnant or breastfeeding individuals.
* Patients with contraindications to ileo-colonoscopy (e.g., severe comorbidities, known intolerance).
* Individuals unable to provide informed consent.
* Patients with conditions interfering with ultrasound imaging, such as severe obesity or uncooperative behaviour

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Mid-End and High-End Ultrasound in Detecting Ileocolonic Inflammation Compared to Ileo-Colonoscopy | Day 1 (same day as colonoscopy)
  Diagnostic accuracy (sensitivity, specificity, positive predictive value, and negative predictive value) of mid-end ultrasound (Siemens ACUSON S2000) and high-end ultrasound (Samsung RS85) in detecting inflammation in the terminal ileum and colon, as compared to findings on ileo-colonoscopy (reference standard). Each patient will undergo both ultrasound examinations followed by ileo-colonoscopy. Sonographic features assessed include bowel wall thickness, mural stratification, and vascularity. Colonoscopy will be scored using validated endoscopic indices such as the Simple Endoscopic Score for Crohn's Disease and the Ulcerative Colitis Endoscopic Index of Severity.

SECONDARY OUTCOMES:
Number of Participants With Change in Clinical Management Based on Ultrasound Findings as Determined by Independent Physician Panel | Within 24 hours of ultrasound examination
  Number of participants in whom treatment decisions (e.g., escalation or de-escalation of medical therapy, surgical referral, or ordering of additional diagnostic testing) were modified based on findings from mid-end or high-end ultrasound. An independent, blinded panel of three inflammatory bowel disease specialists will review clinical scenarios with and without ultrasound results and adjudicate whether ultrasound findings contributed to a management change.

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No